CLINICAL TRIAL: NCT00232063
Title: Long-term Study of Ciclosporin for Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLO400D1304
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Severe Atopic Dermatitis
Keywords: Atopic Dermatitis, Ciclosporin,
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cyclosporine

INTERVENTIONS:
Drug: ciclosporin

SUMMARY:
In patients with severe adult atopic dermatitis, the safety and efficacy of OL27-400MEPC will be assessed by repeating oral administration at a dose of 3 mg/kg/day (2-5 mg/kg/day) in 2 divided doses daily for 8-12 weeks and recovery until 52 weeks after starting treatment

ELIGIBILITY:
Inclusion Criteria:

* - Appropriate the definition/diagnosis criteria of atopic dermatitis of the Japanese Dermatological Association
* Patients with severest atopic dermatitis [according to the "Guidelines for Treatment of Atopic Dermatitis 2002, the severity of atopic dermatitis will be classified as severest when an eruption associated with severe inflammation (a lesion associated with erythema, papule, erosion, infiltration, lichenification, etc.) is noted on at least 30% of body surface on the day of subject enrollment].

Exclusion Criteria:

* Patients who received oral preparations, injections, inhaled preparations and suppositories of steroids or immunosuppressants other than tacrolimus hydrate ointments within 14 days of subject enrollment
* Patients who might receive the oral/injection drugs which are known to enhance nephrotoxicity, increase serum potassium levels, HMG-CoA reductase inhibitors or theophylline during the treatment period.
* Patients who received or are receiving an ultraviolet therapy (PUVA therapy, etc.)
* Patients with hypertension, active infectional disease, gout etc. Other protocol-defined exclusion criteria may apply.

Ages: 20 Years to 64 Years | Sex: All
Age Groups: Adult
Dates: Start 2004-05; Primary Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Japan, Study Chair — Novartis Pharmaceuticals Japan